CLINICAL TRIAL: NCT02624258
Title: Pilot Study of Non-Viral, RNA-Redirected Autologous T Cells Engineered to Contain Anti-CD19 Linked to TCR and 4-1BB Signaling Domains in Patients With Refractory or Relapsed Hodgkin Lymphoma
Brief Title: Pilot Study of Non-Viral, RNA-Redirected Autologous T Cells in Patients With Refractory or Relapsed Hodgkin Lymphoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Principal Investigator decision to stop trial
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14BT055, 821157
Record Dates: First submitted 2015-12-01; First posted 2015-12-08 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RNA CART19 cells (Experimental): CD19 RNA redirected autologous T-cells (RNA CART19 cells)
  Interventions: Biological: CD19 RNA redirected autologous T-cells (RNA CART19 cells)

INTERVENTIONS:
Biological: CD19 RNA redirected autologous T-cells (RNA CART19 cells) — Subjects will be treated with IV administration of RNA anti-CD19 CAR T cells for a total of six doses over 3 weeks. The first dose will be administered 1-4 days after infusion of cyclophosphamide 30mg/kg.

SUMMARY:
Pilot open-label study to estimate the feasibility, safety and efficacy of intravenously administered, RNA electroporated autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ /4-1BB) costimulatory domains (referred to as "RNA CART19") in Hodgkin Lymphoma (HL) patients. Subjects will be treated with IV administration of RNA anti-CD19 CAR T cells for a total of six doses over 3 weeks.

DETAILED DESCRIPTION:
The study will enroll 10 evaluable patients. Evaluable patients are those who have received at least 1 of the 6 RNA CART19 doses at the protocol-specified level. Important safety data can be collected even if a patient receives only one RNA CART19 dose. Subjects (n = 10) will receive up to six IV doses of 8x105-1.5x106 RNA CART19 cells/kg/dose for subjects<80kg and 1x108 RNA CART19 cells/dose (±20%) for subjects ≥80kg.

The RNA CART19 doses and mid-treatment single dose cyclophosphamide will be administered on Mondays, Wednesdays or Fridays. Dosing can be initiated on any of those days. Subjects will be infused in a staggered fashion at two week intervals; that is, the next subject cannot be infused prior to two weeks since the last infusion of the previous subject.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with HL with no available curative treatment options (such as autologous SCT) who have a limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled.

  * HL with biopsy-proven relapse or refractory disease who are unresponsive to or intolerant of at least one line of standard salvage therapy;
  * Patients must have evaluable disease by radiologic imaging (FDG PET-CT or FDG PET-MRI) within 42 day of enrollment; evaluable includes both assessable and/or measurable disease
* Age 18 to 24 years. Patients ages 22-24 will only be enrolled if they are currently being treated at CHOP or another pediatric facility/oncologist.
* Expected survival > 12 weeks at time of screening
* Adequate organ function defined as:
* Renal function defined as:

  * Creatinine clearance or radioisotope GFR > 60 mL/min/1.73 m2 OR
  * Serum creatinine: < 1.7mg/dL (male subjects) or < 1.4mg/dL (female subjects)
* ALT < 5 times the ULN for age
* Total Bilirubin < 2.0 mg/dl
* Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation > 94% on room air
* Patients with relapsed disease after prior allogeneic SCT (myeloablative or non-myeloablative) will be eligible if they meet all other inclusion criteria and
* Have no active GVHD and require no immunosuppression
* Are more than 6 months from transplant 6) Karnofsky performance status ≥ 50 at screening
* Left Ventricular Shortening Fraction (LVSF) > 28% confirmed by echocardiogram, or Left Ventricular Ejection Fraction (LVEF) > 45% confirmed by echocardiogram or MUGA
* Signed written informed consent must be obtained prior to any study procedures
* Successful T cell test expansion (to be performed as part of inclusion criteria until 3 subjects meet all enrollment criteria)

Exclusion Criteria:

* Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum pregnancy test at enrollment. A urine pregnancy test will be performed within 48 hours before the RNA CART19 infusion.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* HIV infection.
* Patients with known active CNS involvement by malignancy. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment
* Patients in complete remission with no evidence by radiologic imaging of disease.
* History of allergy to murine proteins
* History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
* Anti-CD20 monoclonal antibody therapy within the last 3 months, or absence of circulating B cells
* Unstable angina and/or myocardial infarction within 6 months prior to screening.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11; Primary Completion 2019-06-05 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events, defined as NCI CTCAE V4 > Grade 3 | Month 4 post-CART19 Infusion
  Occurrence of study related adverse events, defined as NCI CTCAE V4 > grade 3 signs/symptoms, laboratory toxicities and clinical events that are possible, likely or definitely related to study treatment at any time from the first cyclophosphamide infusion until Month 4.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rheingold, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Svoboda J, Rheingold SR, Gill SI, Grupp SA, Lacey SF, Kulikovskaya I, Suhoski MM, Melenhorst JJ, Loudon B, Mato AR, Nasta SD, Landsburg DJ, Youngman MR, Levine BL, Porter DL, June CH, Schuster SJ. Nonviral RNA chimeric antigen receptor-modified T cells in patients with Hodgkin lymphoma. Blood. 2018 Sep 6;132(10):1022-1026. doi: 10.1182/blood-2018-03-837609. Epub 2018 Jun 20. PMID 29925499